CLINICAL TRIAL: NCT06846580
Title: Role of 2 Stages Brachiobasilic Arteriovenous Fistula in Patients Having Central Venous Stenosis with Exhausted Options of Dialysis Access
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Hussein Hassan Ibrahim, Dr., Assiut University
Other Study IDs: BBAVF with CVS
Record Dates: First submitted 2025-02-13; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Brachiobasilic Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: brachiobasilic AVF — perform 2 stage brachiobasilic AVF in hemodialysis patients with central venous stenosis

SUMMARY:
Central venous stenosis (CVS) is a common problem facing the hemodialysis patients planning to receive dialysis through arteriovenous fistula.

The causes for Central venous stenosis are Subclavian and internal jugular catheters which is related mostly to the frequency and the duration of catheters placement. (5) Also, Smaller caliber central venous catheters (such as peripherally inserted central [PICC] and triple-lumen catheters) can also be associated with thrombus formation and Central venous stenosis over a short term.(6) Pacemakers can be a cause which is associated with a 50% prevalence of subclavian vein stenosis.(7) Subclavian catheter placement is a particularly high risk, with the development of subclavian vein stenosis in approximately 25%-50% of patients in various studies.(8,9) The problem now is there is a hemodialysis patient with exhausted options for AVF and a patent basilic vein but the patient has ipsilateral Central venous stenosis. In previous studies, when creating an AVF over central venous stenosis , the investigators preferred to create a Radiocephalic AVF or Brachiocephalic AVF if Radiocephalic AVF is not available. (10) our study proposing the 2 stage brachiobasilic fistula for patients otherwise have no other option for arteriovenous fistula.

Staging the Brachiobasilic procedure will avoid larger incision with the need for general anesthesia until functioning fistula is ensured and central venous stenosis has been delt with.

DETAILED DESCRIPTION:
Central venous stenosis (CVS) is a common problem facing the hemodialysis patients planning to receive dialysis through arteriovenous fistula. The true incidence and prevalence of Central venous stenosis in the ESRD population is unknown because most studies of Central venous stenosis are limited to symptomatic patients. Central venous stenosis may remain asymptomatic because clinical symptoms and signs of Central venous stenosis often develop only after an AVF is placed in the ipsilateral extremity and the impediment to increased blood flow is unmasked. (1) Retrospective investigations of symptomatic HD patients with various accesses using duplex ultrasonography or angiography have reported Central venous stenosis prevalences of 19%-41%. (2-4) The causes for Central venous stenosis are Subclavian and internal jugular catheters which is related mostly to the frequency and the duration of catheters placement. (5) Also, Smaller caliber central venous catheters (such as peripherally inserted central [PICC] and triple-lumen catheters) can also be associated with thrombus formation and Central venous stenosis over a short term.(6) Pacemakers can be a cause which is associated with a 50% prevalence of subclavian vein stenosis.(7) Subclavian catheter placement is a particularly high risk, with the development of subclavian vein stenosis in approximately 25%-50% of patients in various studies.(8,9) The problem now is there is a hemodialysis patient with exhausted options for AVF and a patent basilic vein but the patient has ipsilateral Central venous stenosis. In previous studies, when creating an AVF over central venous stenosis , the investigators preferred to create a Radiocephalic AVF or Brachiocephalic AVF if Radiocephalic AVF is not available. (10) our study proposing the 2 stage brachiobasilic fistula for patients otherwise have no other option for arteriovenous fistula.

Staging the Brachiobasilic procedure will avoid larger incision with the need for general anesthesia until functioning fistula is ensured and central venous stenosis has been delt with.

our Aims are : Evaluates the efficacy and safety of creation of a Brachiobasilic fistula in hemodialysis patients with central venous stenosis Evaluate the outcomes of Superficialization of the basilic vein after percutaneous transluminal angioplasty of the central venous stenosis

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis patients with asymptomatic central venous stenosis that have only basilic vein feasible for creating AVF in one upper limb with exhausted other options for AVF
* Age > 18
* Patent brachial artery by duplex with PSV > 45 cm/s
* Patent Basilic vein with diameter > 3 mm

Exclusion Criteria:

* Patient with other arteriovenous access options
* Patient not fit for surgery
* Patient with Peripheral arterial disease at Upper limb
* Patient with history of DVT in upper limb
* Hemodynamically unstable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with central venous stenosis with exhausted options of dialysis access that has only basilic vein feasible for creation of the fistula
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success of 1st stage Brachiobasilic fistula | through study completion, an average of 2 year
  Palpable thrill Fistula flow rate with duplex ultrasound
Primary patency | through study completion, an average of 2 year
  It is defined as the interval between initial creation of the fistula and its failing that requires endovascular or surgical intervention.
Assisted primary patency | through study completion, an average of 2 year
  It is defined as the time interval of the fistula remaining patent (functional) with the aid of endovascular intervention.

SECONDARY OUTCOMES:
complications of the fistula | through study completion, an average of 2 year
  Bleeding Infection Thrombosis aneurysm formation Distal limb ischemia Severe venous hypertension.
Fistula maturation | 4 weeks after the fistula creation and every 2 weeks up to 24 weeks
  It is defined as flow through the fistula greater than 600 ml/minute, vein diameter more than 6 mm and the vein less than 6 mm from the skin and adequate urea clearance with dialysis.

REFERENCES:
- [Background] Jennings WC, Maliska CM, Blebea J, Taubman KE. Creating arteriovenous fistulas in patients with chronic central venous obstruction. J Vasc Access. 2016 May 7;17(3):239-42. doi: 10.5301/jva.5000507. Epub 2016 Feb 5. PMID 26847733
- [Background] Agarwal AK. Central vein stenosis: current concepts. Adv Chronic Kidney Dis. 2009 Sep;16(5):360-70. doi: 10.1053/j.ackd.2009.06.003. PMID 19695504
- [Background] Barrett N, Spencer S, McIvor J, Brown EA. Subclavian stenosis: a major complication of subclavian dialysis catheters. Nephrol Dial Transplant. 1988;3(4):423-5. doi: 10.1093/oxfordjournals.ndt.a091691. PMID 3140128
- [Background] Schwab SJ, Quarles LD, Middleton JP, Cohan RH, Saeed M, Dennis VW. Hemodialysis-associated subclavian vein stenosis. Kidney Int. 1988 Jun;33(6):1156-9. doi: 10.1038/ki.1988.124. PMID 2969991
- [Background] Sticherling C, Chough SP, Baker RL, Wasmer K, Oral H, Tada H, Horwood L, Kim MH, Pelosi F, Michaud GF, Strickberger SA, Morady F, Knight BP. Prevalence of central venous occlusion in patients with chronic defibrillator leads. Am Heart J. 2001 May;141(5):813-6. doi: 10.1067/mhj.2001.114195. PMID 11320371
- [Background] Grove JR, Pevec WC. Venous thrombosis related to peripherally inserted central catheters. J Vasc Interv Radiol. 2000 Jul-Aug;11(7):837-40. doi: 10.1016/s1051-0443(07)61797-7. PMID 10928518
- [Background] Agarwal AK. Central vein stenosis. Am J Kidney Dis. 2013 Jun;61(6):1001-15. doi: 10.1053/j.ajkd.2012.10.024. Epub 2013 Jan 3. PMID 23291234
- [Background] MacRae JM, Ahmed A, Johnson N, Levin A, Kiaii M. Central vein stenosis: a common problem in patients on hemodialysis. ASAIO J. 2005 Jan-Feb;51(1):77-81. doi: 10.1097/01.mat.0000151921.95165.1e. PMID 15745139
- [Background] Clark DD, Albina JE, Chazan JA. Subclavian vein stenosis and thrombosis: a potential serious complication in chronic hemodialysis patients. Am J Kidney Dis. 1990 Mar;15(3):265-8. doi: 10.1016/s0272-6386(12)80772-4. PMID 2305766
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26847733/